CLINICAL TRIAL: NCT06766461
Title: Beta-Lactam Antibiotics InitiaL ExpoSure OptimisEd in CriticallY Ill Patients with SEpsis
Acronym: BULLSEYE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Maasstad Hospital (Other); Albert Schweitzer Hospital (Other)
Responsible Party: Principal Investigator, Birgit Koch, Principal Investigator, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-512950-13; 10140022310046 (Other Grant/Funding Number: ZonMW); 2024-512950-13-00 (EU CTIS Number); U1111-1308-9223 (Registry Identifier: WHO universal trial number (UTN))
Record Dates: First submitted 2024-11-27; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Sepsis - to Reduce Mortality in the Intensive Care Unit; Sepsis; Septic Shock
Keywords: sepsis; intensive care; critically ill; antibiotic; septic shock
MeSH Terms: conditions — Sepsis; Shock, Septic; Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): This arm will receive standard of care according to local protocol.
- Intervention (Experimental): This arm will be treated with double dosages of beta-lactam antibiotics the first 48 hours after inclusion.
  Interventions: Drug: Double dosing of beta-lactam antibiotic

INTERVENTIONS:
Drug: Double dosing of beta-lactam antibiotic — This arm will receive double dosing of beta-lactam antibiotics for the first 48 hours after inclusion.
  Arms: Intervention

SUMMARY:
The aim of this study is to investigate if an initial short double dose of beta-lactam antibiotics will reduce mortality in critically ill patients with sepsis.

DETAILED DESCRIPTION:
Objective

To determine if using higher dosages of beta-lactam antibiotics in the initial phase of sepsis improves clinical outcome of critically ill patients.

Main trial endpoints

The main trial endpoint is all cause 28-day mortality.

Secondary trial endpoints

Secondary trial endpoints include: Hospital length of stay, ICU length of stay, microbiological eradication, time to shock reversal, clinical cure, Δ Lactate, Δ PCT, Δ SOFA, 90- day mortality, 365-day mortality, pharmacodynamic target, post study calculation of the costs in both study, groups, EQ5D questionnaire 3 and 12 months after Admission, iMTA productivity questionnaire 3 and 12 months after admission, iMTA medical consumption questionnaire 3 and 12 months after admission and the number of adverse events.

Trial design

This is an open label, randomized controlled trial.

Trial population

The trial population will consist of adult patients admitted to the intensive care department with sepsis who will be treated according to protocol with beta-lactam antibiotics.

Interventions

During the trial participants in the intervention group will receive a double dose of antibiotics for the first 48 hours in comparison to the standard dose in the control group.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Receiving intravenous antibiotic therapy of the target drugs (including continuous infusion of beta-lactam antibiotics)
* Primary infection
* Admitted to the ICU
* Meeting the Sepsis-3 criteria for septic shock: sepsis in addition to shock requiring the start of vasopressors to maintain a mean arterial pressure 65 mmHg or greater, and a serum lac tate level greater than 2.0 mmol/L following "adequate fluid resuscitation".

Exclusion Criteria:

* Patient or legal representative not available to give informed consent within 72 hours after admittance
* Pregnancy
* Admittance for burn wounds
* Patients receiving target antibiotics only as prophylaxis within the context of Selective Diges tive tract Decontamination (SDD)
* Enrolment in another interventional trial
* Patient received the study antibiotic for more than 24 hours before inclusion
* Patient receiving extracorporeal membrane oxygenation (ECMO)
* Patient is already treated with a double dose of antibiotics based on suspected infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 980 (Estimated)
Dates: Start 2025-01-03 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
28-day mortality | From enrollment to 28 days

SECONDARY OUTCOMES:
90-day mortality | From enrollment to 90 days
365-day mortality | From enrollment to the 365 days
ICU lengt of stay | From enrollment to the end of the study period at 12 months
Hospital lengt of stay | From enrollment to the end of the study period at 12 months
Time to shock reversal | From enrollment to the end of the study period at 12 months
  From enrollment to the use of <0.1 gamma of vasopressors for 4 consecutive hours.
Microbiological eradication | From enrollment to hospital discharge
  Eradication of the causative organism from the primary source up to 30 days after therapy when confirmed by at least one repeated culture. In cases where there were no repeat cultures and the patient had resolution of the infection, microbial eradication will be presumed.
Clinical cure | From enrollment to 14 days
  Completion of β-lactam antibiotic by day 14 without recommencement of antibiotics within 48hrs of cessation for same infective episode (investigator assessment of clinical response)
Plasma concentrations of the beta-lactam antibiotics | From enrollment to day 3
  Through concentrations take once a day for 3 consectutive days after enrollment. Target attianment is defined as 100%fT>4xMIC
Delta SOFA | From enrollment to day 3
  SOFA at day 3 - SOFA at admission
Delta Lactate | From enrollment to day 3
  Lactate at day 3 - lactate upon inclusion
Quality of life | 3 and 12 months after inclusion
  EQ-5D-5L, a quetionnaire scoring 1 to 5 points on 5 domains. A higher score means a worse outcome.
Medical consumption | 3 and 12 months after inclusion
  iMTA Medical Consumption questionnaire
Productivity | 3 and 12 months after inclusion
  iMTA Productivity questionnaire
Adverse events and toxicity | From enrollment until the end of the study period at 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Maasstad Ziekenhuis, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Horstink MMB, Geel DR, den Uil CA, Deetman PE, Endeman H, Abdulla A, Bosch TM, Rietdijk WJR, Thielen FW, Haringman JJ, van Vliet P, Rijpstra TA, Bethlehem C, Beishuizen A, Muller AE, Koch BCP; BULLSEYE investigators. Standard versus double dosing of beta-lactam antibiotics in critically ill patients with sepsis: The BULLSEYE study protocol for a multicenter randomized controlled trial. BMC Infect Dis. 2025 Mar 21;25(1):392. doi: 10.1186/s12879-025-10747-3. PMID 40119275